CLINICAL TRIAL: NCT03068156
Title: Efficacy of 308-nm Excimer Laser for Primary Localized Cutaneous Amyloidosis Treatment in Asians: Pilot Study
Brief Title: Efficacy of 308-nm Excimer Laser for Primary Localized Cutaneous Amyloidosis Treatment in Asians
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Collaborators: Ratchadapiseksompotch Fund (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CU_308excimer_amyloidosis
Record Dates: First submitted 2017-02-20; First posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Lichen Amyloidosis
Keywords: 308-nm excimer laser; primary localized cutaneous amyloidosis; lichen amyloidosis; Asians
MeSH Terms: conditions — Amyloidosis, Primary Cutaneous | interventions — Lasers, Excimer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- excimer laser (Experimental)
  Interventions: Radiation: 308-nm excimer laser
- Control (No Intervention)

INTERVENTIONS:
Radiation: 308-nm excimer laser — monochromator UVB laser (308nm)
  Arms: excimer laser

SUMMARY:
Efficacy of 308-nm excimer laser for primary localized cutaneous amyloidosis treatment in Asians, pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Patients, aged >18 years old with lichen amyloidosis diagnosed by using clinical presentation and pathologic features

Exclusion Criteria:

* Those with cutaneous amyloidosis associated systemic diseases
* Pregnancy or lactating woman
* Those who are allergic to urea, olive oil
* Those who are photosensitive to ultraviolet radiation
* Those who had been previously treated with medications/ radiation/ laser within 3 months for systemic and 1 month for topical therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-01-31 (Actual); Primary Completion 2018-01-30 (Estimated); Study Completion 2018-03-02 (Estimated)

PRIMARY OUTCOMES:
Roughness evaluation by using Visioscan® VC98 | Change from baseline roughness at every 2 weeks up to 16 weeks
  The improvement of roughness evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Einapak Amnarttrakul, M.D., Principal Investigator — Chulalongkorn University
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided